CLINICAL TRIAL: NCT02617459
Title: A Multicenter, Randomized, Open-label, Positive-controlled, Parallel-group Clinical Trial of Levobetaxolol Hydrochloride Eye Drops in Patients With Primary Open-angle Glaucoma or Ocular Hypertension
Brief Title: Levobetaxolol Hydrochloride Eye Drops for Treatment of Primary Open-angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZK-LBL-2016-01
Record Dates: First submitted 2015-11-18; First posted 2015-12-01 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Primary Open-angle Glaucoma; Ocular Hypertension
Keywords: Safety; efficacy; Levobetaxolol eye drops; Chinese patients
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levobetaxolol eye drops (Experimental): Levobetaxolol eye drops 5ml/25mg per bottle
  Interventions: Drug: Levobetaxolol eye drops
- Betaxolol eye drops (Active Comparator): Betaxolol eye drops 5ml/12.5mg per bottle
  Interventions: Drug: Betaxolol eye drops

INTERVENTIONS:
Drug: Levobetaxolol eye drops — one drop per time; twice daily
  Arms: Levobetaxolol eye drops
Drug: Betaxolol eye drops — one drop per time; twice daily
  Arms: Betaxolol eye drops

SUMMARY:
To evaluate the safety and efficacy of Levobetaxolol in Chinese patients with glaucoma.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of Levobetaxolol in Chinese patients with primary open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Agreed to participate in this clinical trial and informed consent;
* Aged 18 to 70 years of age, male or female;
* In line with primary open-angle glaucoma diagnostic criteria, IOP ≥18mmHg;
* or in compliance with ocular hypertension diagnostic criteria, intraocular pressure> 21mmHg

Exclusion Criteria:

* Known or suspected to be allergic to investigational drugs and materials
* has been diagnosed with angle-closure glaucoma, absolute glaucoma, glaucoma ciliary body syndrome, secondary glaucoma.
* merge various retinal lesions, such as retinal detachment, retinal vein occlusion, retinitis pigmentosa.
* merge associated with eye infections or cornea, iris, lens obvious lesions, or one-eyed patients.
* During the trial who must wear contact lenses, or nearly three months experts any eye surgery or laser treatment.
* Need systemic β-blocker therapy during the study.
* with severe kidney disease, or abnormal liver function tests (ALT, AST≥ 1.5 times the upper limit of normal, SCr> upper limit of normal).
* merge sinus bradycardia, over Ⅰ degree atrioventricular block, cardiogenic shock, heart failure, symptomatic hypotension or other serious heart, lung diseases (such as bronchial asthma or a history of bronchial asthma, chronic obstructive lung disease, bronchospasm, respiratory failure, etc.).
* merge hyperthyroidism, myasthenia gravis, diabetes, advanced cancer, blood and hematopoietic system diseases, or other serious or progressive disease systems.
* associated with neurological and psychiatric disorders
* suspect or indeed alcohol, drug abuse history.
* pregnancy, lactation or recent fertility planner.
* The researchers believe other circumstances were not involved in this trial.
* participate in other clinical trials within three months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Change in intraocular pressure (IOP) from baseline at week 8 after the treatment (a.m.) | 8 weeks
  Change in intraocular pressure (IOP) from baseline at week 8 after the treatment (a.m.)

SECONDARY OUTCOMES:
Change in intraocular pressure (IOP) from baseline to week 2 | 2 weeks
  Change in intraocular pressure (IOP) from baseline to week 2
Change in intraocular pressure (IOP) from baseline to week 4 | 4 weeks
  Change in intraocular pressure (IOP) from baseline to week 4
Change in intraocular pressure (IOP) from baseline to week 8 (p.m.) | 8 weeks
  Change in intraocular pressure (IOP) from baseline to week 8 (p.m.)
Change from baseline in mean visual field defect (MD) at 8 weeks after the treatment | 8 weeks
  Change from baseline in mean visual field defect (MD) at 8 weeks after the treatment
Change in visual field pattern standard deviation (PSD) from baseline at 8 weeks after the treatment | 8 weeks
  Change in visual field pattern standard deviation (PSD) from baseline at 8 weeks after the treatment
Change in retinal nerve fiber layer (RNFL) thickness from baseline at 8 weeks after the treatment | 8 weeks
  Change in retinal nerve fiber layer (RNFL) thickness from baseline at 8 weeks after the treatment
Change in visual acuity test at week 2 | 2 weeks
  Change in visual acuity test at week 2
Change in visual acuity test at week 4 | 4 weeks
  Change in visual acuity test at week 4
Change in visual acuity test at week 8 | 8 weeks
  Change in visual acuity test at week 8

CONTACTS AND LOCATIONS:
Overall Officials: Jian Ge, MD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan ophthalmic center, Sun Yat-sen University, Guangzhou, Guangdong, China